CLINICAL TRIAL: NCT04018638
Title: B-FREE in the UP! Improving Recovery After a Knee Replacement With Blood-Flow Restriction Exercise Enhancement
Brief Title: Blood-Flow Restriction Exercise Following a Knee Replacement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan Technological University (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MichiganTU
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Knee Injuries; Knee Osteoarthritis; Knee Arthritis
MeSH Terms: conditions — Knee Injuries; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adults with TKR Perform Home Exercise Program (Experimental): Participants that have a total knee replacement will complete a home-based exercise program
  Interventions: Other: B-FREE
- Healthy Controls Only (No Intervention): Participants that have no history of knee joint dysfunction will serve as age-matched uninjured controls

INTERVENTIONS:
Other: B-FREE — Blood flow-restriction exercise enhancement (B-FREE) will be performed at home 3x/wk for 10 weeks. A blood pressure cuff will be inflated to partially occlude blood to the limb during light weight exercises involving knee extension, body weight squats, and walking.
  Arms: Adults with TKR Perform Home Exercise Program

SUMMARY:
This study will determine the safety and efficacy of using blood-flow restriction exercise enhancement (B-FREE) to overcome persistent quadriceps muscle weakness that occurs following a total knee replacement (TKR).

DETAILED DESCRIPTION:
This study aims to determine the safety and efficacy of using B-FREE to overcome persistent quadriceps muscle weakness that occurs following a TKR. We hypothesize that B-FREE can provide a safe training stimulus and offer a home-based program to restore quadriceps muscle strength and improve functional mobility. Specifically, subjects that have a TKR will perform B-FREE at home (light weights with resistance bands and walking) 3x/wk for 10 weeks. Quadriceps muscle strength, balance, and functional mobility will be assessed before and after the program. Changes in these variables will be compared to healthy age-matched uninjured controls.

ELIGIBILITY:
Inclusion Criteria

* 40-75 years of age
* Have had a unilateral TKA > 6 months prior to participation (Arm 1)
* No previous history of knee injury/surgery (Arm 2)

Exclusion Criteria

* Are a smoker
* Have diabetes
* Have suffered a heart attack or stroke
* Have any cardiopulmonary disorders (hypertension discussed below)
* Have been diagnosed with any neurological disorders
* Have any implanted devices such as but not limited to a pacemaker or pain pump
* Uncontrolled (not medicated) Stage 1 hypertension or Stage 2 hypertension

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle size | Change from baseline at 10 weeks
  quadriceps muscle thickness
Change in Muscle strength | Change from baseline at 10 weeks
  quadriceps muscle strength

SECONDARY OUTCOMES:
Change in Walking performance | Change from baseline at 10 weeks
  walking distance
Change in Balance | Change from baseline at 10 weeks
  balance assessment

CONTACTS AND LOCATIONS:
Overall Officials: Steven Elmer, Principal Investigator — Michigan Technological University
Locations (1):
- Michigan Technological University, Houghton, Michigan, United States

IPD SHARING:
Plan to Share IPD: No